CLINICAL TRIAL: NCT06676462
Title: Pilot Study Comparing the HEINE visionPRO HyMac 3 and the GlideScope Hyperangulated S3 Laryngoscope Blade on Time to Intubation
Brief Title: Non-inferiority Trial Comparing visionPRO to Glidescope Video Laryngoscopes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ruediger Noppens, Anesthesiologist, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: visionPRO vs. Glidescope
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication; Video Laryngoscopy; Airway Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video laryngoscopy with visionPRO (Experimental): Video laryngoscopy will be performed with the visionPRO (HEINE® Optotechnick, Gilching, Germany)
  Interventions: Device: Video laryngoscopy with visionPRO
- Video laryngoscopy with Glidescope (Active Comparator): Video laryngoscopy will be performed with the GlideScope (Verathon Inc., Bothell, USA)
  Interventions: Device: Video laryngoscopy with Glidescope

INTERVENTIONS:
Device: Video laryngoscopy with visionPRO — Video laryngoscopy to be performed using the visionPRO (HEINE® Optotechnick, Gilching, Germany) during intubation.
  Arms: Video laryngoscopy with visionPRO
Device: Video laryngoscopy with Glidescope — Video laryngoscopy to be performed using theGlideScope (Verathon Inc., Bothell, USA) during intubation.
  Arms: Video laryngoscopy with Glidescope

SUMMARY:
Indirect video laryngoscope tracheal intubation with the GlideScope (Verathon Inc., Bothell, USA) has become a well-established technique in emergency and clinical anaesthesia, offering first-pass intubation success rates comparable to those achieved with direct laryngoscopy. Different video laryngoscopes vary significantly in design, including blade shape, mobility, and camera operation, which can affect patient outcomes. Two video laryngoscopes with hyperangulated blades include the GlideScope (Verathon Inc., Bothell, USA) and the visionPRO (HEINE® Optotechnick, Gilching, Germany). The Glidescope comprises an external monitor connected to a medical-grade plastic handle which is compatible with reusable and disposable blades. The newer visionPro comprises a reusable anodized aluminum integrated monitor that is attached to the camera/handle which is compatible with disposable blades. The hyperangulated blade of the VisionPro is a unique combination of previously designed laryngoscope blades meant to increase performance. The introduction of this new hyperangulated blade design in the VisionPro raises the need to compare its performance against the established GlideScope.

The aim of this pilot study is to generate initial data to evaluate whether the use of the visionPRO (HEINE® Optotechnick, Gilching, Germany) provides a non-inferior first-pass success rate compared with the GlideScope (Verathon Inc., Bothell, USA) in surgical patients with an expected normal airway undergoing general anaesthesia The investigators hypothesize that tracheal intubation using the HEINE visionPRO will achieve a similar frequency of failed intubation and airway complications. This study plans to recruit 100 patients.

DETAILED DESCRIPTION:
This trial is a single-centre, pilot, patient-blinded, randomized controlled non-inferiority trial.

Patients who decide to participate in this study will have their surgery and follow up care proceed according to standard of care. Video laryngoscopy is standard of care for this patient population at LHSC. Once eligibility is confirmed and informed, written consent has been obtained, participants be randomized to one of two study groups:

1. Laryngoscopy performed using the Glidescope device (Verathon Inc., Bothell, USA)
2. Laryngoscopy performed using the visionPRO device (HEINE® Optotechnick, Gilching, Germany)

Surgery, anesthetic management, and intubation protocol will proceed according to standard of care.

(A) All patients are observed for ECG, oxygen saturation (SpO2), and non-invasive blood pressure. Pre-oxygenation is carried out by the provider based on patient characteristics and standard clinical procedures (EtO2 > 80%).

(B) After adequate pre-oxygenation, anaesthesia is initiated using a combination of fentanyl (0.1 - 0.15 µg.kg-1) / sufentanil (0.2 - 0.5 µg.kg-1), and propofol (2 - 3 mg.kg-1), with the choice of drugs and dosages tailored to the specific needs of the patient. Maintenance is achieved either through propofol infusion (TIVA) or inhaled anaesthetics. The selection of a neuromuscular blocking agent is based on the surgery's duration, the need for perioperative neurological monitoring, and the absence of allergies and organ failures. The agents and their dosages used are:

1. Rocuronium (0.5 - 1.2 mg.kg-1); and
2. Succinylcholine (1 - 2 mg.kg-1).

The train-of-four (TOF) method is employed by the study nurse for continuous quantitative monitoring of neuromuscular transmission. Complete muscle relaxation is confirmed by the absence of tactile and measured twitches in response to maximal TOF stimulation of the ulnar nerve at the adductor pollicis. Study personnel were instructed on the importance of achieving adequate neuromuscular blockade.

(C) The laryngoscopy attempt starts with a TOF count of 0/4, using the device specified by randomization:

1. visionPRO (HEINE® Optotechnick, Gilching, Germany) or
2. GlideScope (Verathon Inc., Bothell, USA)

The provider aims to achieve the clearest view of the laryngeal structures. External laryngeal manipulations (ELM) may be employed to enhance the view of the glottis, aiming for a Cormack and Lehane grade I or II. The endotracheal tube size and blade size are chosen according to the hospital's standard operating procedures (blade size: #3 for average patients, #4 for taller patients; standard ET sizes: 7.0-7.5 ID for female patients and 7.5-8.0 ID for male patients). The method of glottic visualization and the size of the ET and blade are documented in the case report form (CRF).

(D) An intubation attempt is defined as the insertion and removal of the laryngoscope blade from the mouth, regardless of ET insertion success. A laryngoscopy attempt is considered successful if the tracheal tube is placed with a single blade insertion within 120 seconds and without manipulation of the laryngoscope by another provider. The following times periods until final ET placement are measured by a study nurse via a timer:

1. "Time to intubation": duration from the opening of the patient's mouth to the passage of the ET through the vocal cords.
2. "Time to view": the time from device insertion to visualization of the glottis;
3. "Time to ventilation": the time from device insertion into the mouth until confirmation of the first CO2 wave on the anaesthesia respirator.

If the first attempt fails, the provider makes a second attempt with the same device, with mask ventilation recommended between attempts. A maximum of two laryngoscopy attempts are allowed. After two attempts the clinician switches to a preferred technique and records the direct and/or screen view. If this preferred technique fails after two attempts, the clinician proceeds with a preferred rescue technique. The study protocol recommends this limit of two intubation attempts and alternative technique selection in line with clinical standards. If ELM techniques, such as BURP (specific pressure applied to the cricoid cartilage), are needed during laryngoscopy, they are documented in the CRF. Throughout the induction of anaesthesia, a study nurse not involved in patient care records the study parameters.

24 hours following surgery, the patient will be assessed for presence and severity of sore throat rated on a scale of 0-3 (0 meaning no sore throat and 3 meaning severe sore throat), hoarseness rated on a scale of 0-3 (0 meaning no complaint and 3 meaning severe hoarseness), and cough rated on a scale of 0-3 (0 meaning no cough and 3 meaning severe cough).

ELIGIBILITY:
Inclusion Criteria:

* Having elective surgery with general anesthesia
* At least 18 years of age
* requiring mechanical ventilation via an oral endotracheal tube

Exclusion Criteria:

* More than one predictor of an anticipated difficult airway (eg, body mass index (BMI) >40 kg/m2, unanticipated difficult airway in the medical history (eg, Cormack & Lehane (C&L) ≥III), reduction of the atlanto-occipital joint extension <35°, reduced thyromental distance <6 cm or Mallampati class ≥III)
* Age <18 years
* ASA class IV-VI
* Pregnant or breastfeeding
* Unable to provide informed written consent or under guardianship
* Urgent surgical intervention
* At high risk for aspiration
* Patients undergoing any neck and throat surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Initial or first-pass success rate of indirect video laryngoscope endotracheal intubation (ET) | 0-120 seconds for first pass intubation attempt.
  The primary outcome compares the initial or first-pass success rate of indirect video laryngoscope endotracheal intubation (ET) with the HyMac blade of the visionPRO (HEINE® Optotechnick, Gilching, Germany) to the hyperangulated blade of the GlideScope (Verathon Inc., Bothell, USA) in patients undergoing elective surgery and requiring tracheal intubation. This will be measured by recording how long it takes for successful intubation to take place using the above-mentioned devices, and any complications that may have arisen during the intubation procedure.

SECONDARY OUTCOMES:
Incidence and severity of patient-reported postoperative sore throat (POST) during the first 24 hours | 24 hours following surgery
  The secondary outcome compares the incidence and severity of patient-reported postoperative sore throat (POST) during the first 24 hours. This will be measured by asking patients to rate any occurrence of sore throat on a scale of 0-3 (0 meaning no sore throat and 3 meaning severe sore throat) 24 hours following surgery

OTHER OUTCOMES:
Timing of tracheal intubation events | Duration of intubation procedure
  1. "Time to intubation": duration from the opening of the patient's mouth to the passage of the ET through the vocal cords.
  2. "Time to view": the time from device insertion to visualization of the glottis.
  3. "Time to ventilation": the time from device insertion into the mouth until confirmation of the first CO2 wave on the anaesthesia respirator.
  Measured by recording intubation observations and details during surgery.
Number of laryngoscopy attempts | Duration of intubation procedure
  Number of laryngoscopy attempts required to achieve successful intubation. Measured by recording the number of intubation attempts needed before procedure is successfully executed.
Number of additional operators | Duration of intubation procedure
  Number of operators required to facilitate successful intubation.
  Measured by recording the operators that needed to be involved before procedure is successfully executed.
Lifting force required | Duration of intubation procedure
  Lifting force required (normal or increased) to facilitate successful intubation.
  Measured by recording the physical effort required during laryngoscopy.
Failures/crossovers to other rescue techniques | Duration of intubation procedure
  Instances that intubation failed, required use of other techniques/devices other than the study group (laryngoscopy with either the visionPRO or Glidscope device) the participant was randomized to, or required rescue technique to successfully intubate the patient.
  Measured by recording intubation observations and details during surgery.
Use of extra laryngeal manipulation | Duration of intubation procedure
  Use of extra laryngeal manipulation (applied or not applied) required to complete successful intubation. Measured by recording intubation observations and details during surgery.
Visualization of glottic view | Duration of intubation procedure
  Assessment of glottic view using Cormack and Lehane grading and percentage of glottic opening (POGO) score.
Intubation difficulty | Completion of intubation procedure
  Difficulty of intubation will be assessed using the Intubation Difficulty Score.
Correlation between clinical experiences in airway management and level of training with success rates | Duration of intubation procedure
  Intubation success rates will be correlated to operator experience in anesthesia (consultant or resident and years holding each designation) and experience each operator had performing video laryngoscopy, and comparing this to the details of their intubation attempts.
Complications | Time of surgery to 24 hours postoperative
  Complications for each participant, if applicable (such as desaturation, dental injury, lip injury, glottis injury, other) will be recorded to determine if there is a correlation between complications and video laryngoscope used (visionPRO or Glidescope).
Degree of ease or difficulty of tracheal intubation | Duration of intubation procedure
  Degree of ease or difficulty of tracheal intubation will be measured using a Likert scale (0=easy to 10=difficult) to assess operator-reported difficulty using the video laryngoscopes.
Position of the vocal chords | Duration of intubation procedure
  Positioning of the vocal cords (abducted or adducted) will be assess for each intubation performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ruediger Noppens, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kriege M, Noppens RR, Turkstra T, Payne S, Kunitz O, Tzanova I, Schmidtmann I; EMMA Trial Investigators Group. A multicentre randomised controlled trial of the McGrath Mac videolaryngoscope versus conventional laryngoscopy. Anaesthesia. 2023 Jun;78(6):722-729. doi: 10.1111/anae.15985. Epub 2023 Mar 16. PMID 36928625
- [Background] Yeatts DJ, Dutton RP, Hu PF, Chang YW, Brown CH, Chen H, Grissom TE, Kufera JA, Scalea TM. Effect of video laryngoscopy on trauma patient survival: a randomized controlled trial. J Trauma Acute Care Surg. 2013 Aug;75(2):212-9. doi: 10.1097/TA.0b013e318293103d. PMID 23823612
- [Background] Aziz MF, Healy D, Kheterpal S, Fu RF, Dillman D, Brambrink AM. Routine clinical practice effectiveness of the Glidescope in difficult airway management: an analysis of 2,004 Glidescope intubations, complications, and failures from two institutions. Anesthesiology. 2011 Jan;114(1):34-41. doi: 10.1097/ALN.0b013e3182023eb7. PMID 21150569
- [Background] Ruetzler K, Bustamante S, Schmidt MT, Almonacid-Cardenas F, Duncan A, Bauer A, Turan A, Skubas NJ, Sessler DI; Collaborative VLS Trial Group. Video Laryngoscopy vs Direct Laryngoscopy for Endotracheal Intubation in the Operating Room: A Cluster Randomized Clinical Trial. JAMA. 2024 Apr 16;331(15):1279-1286. doi: 10.1001/jama.2024.0762. PMID 38497992
- [Background] Noppens RR, Mobus S, Heid F, Schmidtmann I, Werner C, Piepho T. Evaluation of the McGrath Series 5 videolaryngoscope after failed direct laryngoscopy. Anaesthesia. 2010 Jul;65(7):716-20. doi: 10.1111/j.1365-2044.2010.06388.x. Epub 2010 Jun 7. PMID 20528841
- [Background] Kaplan A, Goksu E, Yildiz G, Kilic T. Comparison of the C-MAC Videolaryngoscope and Rigid Fiberscope with Direct Laryngoscopy in Easy and Difficult Airway Scenarios: A Manikin Study. J Emerg Med. 2016 Mar;50(3):e107-14. doi: 10.1016/j.jemermed.2015.06.070. Epub 2015 Dec 22. PMID 26725922
- [Background] Savoldelli GL, Schiffer E, Abegg C, Baeriswyl V, Clergue F, Waeber JL. Learning curves of the Glidescope, the McGrath and the Airtraq laryngoscopes: a manikin study. Eur J Anaesthesiol. 2009 Jul;26(7):554-8. doi: 10.1097/eja.0b013e3283269ff4. PMID 19522050
- [Background] Sakles JC, Javedani PP, Chase E, Garst-Orozco J, Guillen-Rodriguez JM, Stolz U. The use of a video laryngoscope by emergency medicine residents is associated with a reduction in esophageal intubations in the emergency department. Acad Emerg Med. 2015 Jun;22(6):700-7. doi: 10.1111/acem.12674. Epub 2015 May 20. PMID 25996773
- [Background] Hasegawa K, Shigemitsu K, Hagiwara Y, Chiba T, Watase H, Brown CA 3rd, Brown DF; Japanese Emergency Medicine Research Alliance Investigators. Association between repeated intubation attempts and adverse events in emergency departments: an analysis of a multicenter prospective observational study. Ann Emerg Med. 2012 Dec;60(6):749-754.e2. doi: 10.1016/j.annemergmed.2012.04.005. Epub 2012 Apr 28. PMID 22542734
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Law JA, Duggan LV, Asselin M, Baker P, Crosby E, Downey A, Hung OR, Jones PM, Lemay F, Noppens R, Parotto M, Preston R, Sowers N, Sparrow K, Turkstra TP, Wong DT, Kovacs G; Canadian Airway Focus Group. Canadian Airway Focus Group updated consensus-based recommendations for management of the difficult airway: part 1. Difficult airway management encountered in an unconscious patient. Can J Anaesth. 2021 Sep;68(9):1373-1404. doi: 10.1007/s12630-021-02007-0. Epub 2021 Jun 18. PMID 34143394
- [Background] Law JA, Duggan LV, Asselin M, Baker P, Crosby E, Downey A, Hung OR, Kovacs G, Lemay F, Noppens R, Parotto M, Preston R, Sowers N, Sparrow K, Turkstra TP, Wong DT, Jones PM; Canadian Airway Focus Group. Canadian Airway Focus Group updated consensus-based recommendations for management of the difficult airway: part 2. Planning and implementing safe management of the patient with an anticipated difficult airway. Can J Anaesth. 2021 Sep;68(9):1405-1436. doi: 10.1007/s12630-021-02008-z. Epub 2021 Jun 8. PMID 34105065
- [Background] Hansel J, Rogers AM, Lewis SR, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adults undergoing tracheal intubation. Cochrane Database Syst Rev. 2022 Apr 4;4(4):CD011136. doi: 10.1002/14651858.CD011136.pub3. PMID 35373840
- [Background] Hansel J, Rogers AM. Mirror, mirror, on the wall, which is the best videolaryngoscope of them all? Anaesthesia. 2022 Apr;77(4):493. doi: 10.1111/anae.15654. Epub 2021 Dec 26. No abstract available. PMID 34957546
- [Background] de Carvalho CC, da Silva DM, Lemos VM, Dos Santos TGB, Agra IC, Pinto GM, Ramos IB, Costa YSC, Santos Neto JM. Videolaryngoscopy vs. direct Macintosh laryngoscopy in tracheal intubation in adults: a ranking systematic review and network meta-analysis. Anaesthesia. 2022 Mar;77(3):326-338. doi: 10.1111/anae.15626. Epub 2021 Dec 1. PMID 34855986
- [Background] Wunsch VA, Kohl V, Breitfeld P, Bauer M, Sasu PB, Siebert HK, Dankert A, Stark M, Zollner C, Petzoldt M. Hyperangulated blades or direct epiglottis lifting to optimize glottis visualization in difficult Macintosh videolaryngoscopy: a non-inferiority analysis of a prospective observational study. Front Med (Lausanne). 2023 Nov 30;10:1292056. doi: 10.3389/fmed.2023.1292056. eCollection 2023. PMID 38098848
- [Background] Kohl V, Wunsch VA, Muller MC, Sasu PB, Dohrmann T, Peters T, Tolkmitt J, Dankert A, Krause L, Zollner C, Petzoldt M. Hyperangulated vs. Macintosh videolaryngoscopy in adults with anticipated difficult airway management: a randomised controlled trial. Anaesthesia. 2024 Sep;79(9):957-966. doi: 10.1111/anae.16326. Epub 2024 May 24. PMID 38789407
- [Background] de Carvalho CC. Hyperangulated vs. Macintosh videolaryngoscopes for efficacy of orotracheal intubation in adults: a pairwise meta-analysis of randomised clinical trials. Anaesthesia. 2022 Oct;77(10):1172-1174. doi: 10.1111/anae.15810. Epub 2022 Jul 21. No abstract available. PMID 35864594
- [Background] Rai MR, Dering A, Verghese C. The Glidescope system: a clinical assessment of performance. Anaesthesia. 2005 Jan;60(1):60-4. doi: 10.1111/j.1365-2044.2004.04013.x. PMID 15601274
- [Background] Fuller RG, Rossetto MA, Paulson MW, April MD, Ginde AA, Bebarta VS, Flarity KM, Keenan S, Schauer SG. Market Analysis of Video Laryngoscopy Equipment for the Role 1 Setting. Mil Med. 2023 Nov 3;188(11-12):e3482-e3487. doi: 10.1093/milmed/usad189. PMID 37338293
- [Background] McCoy EP, Mirakhur RK. The levering laryngoscope. Anaesthesia. 1993 Jun;48(6):516-9. doi: 10.1111/j.1365-2044.1993.tb07075.x. PMID 8292132
- [Background] Nandakumar KP, Bhalla AP, Pandey RK, Baidya DK, Subramaniam R, Kashyap L. Comparison of Macintosh, McCoy, and Glidescope video laryngoscope for intubation in morbidly obese patients: Randomized controlled trial. Saudi J Anaesth. 2018 Jul-Sep;12(3):433-439. doi: 10.4103/sja.SJA_754_17. PMID 30100843
- [Background] Nair SM, Menon GD, George M, Issac E, Bhaskaran R. Comparison of performance characteristics of C-MAC video, McCoy, and Macintosh laryngoscopes in elective cervical spine surgery. J Anaesthesiol Clin Pharmacol. 2021 Oct-Dec;37(4):569-573. doi: 10.4103/joacp.JOACP_56_20. Epub 2022 Jan 6. PMID 35340959
- [Background] Lee SH, Lee YC, Lee JH, Choi SR, Lee SC, Lee JH, Chung CJ. The prophylactic effect of dexamethasone on postoperative sore throat in prone position surgery. Korean J Anesthesiol. 2016 Jun;69(3):255-61. doi: 10.4097/kjae.2016.69.3.255. Epub 2016 Jun 1. PMID 27274371
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Kriege M, Alflen C, Tzanova I, Schmidtmann I, Piepho T, Noppens RR. Evaluation of the McGrath MAC and Macintosh laryngoscope for tracheal intubation in 2000 patients undergoing general anaesthesia: the randomised multicentre EMMA trial study protocol. BMJ Open. 2017 Aug 21;7(8):e016907. doi: 10.1136/bmjopen-2017-016907. PMID 28827261
- [Background] Aziz MF, Abrons RO, Cattano D, Bayman EO, Swanson DE, Hagberg CA, Todd MM, Brambrink AM. First-Attempt Intubation Success of Video Laryngoscopy in Patients with Anticipated Difficult Direct Laryngoscopy: A Multicenter Randomized Controlled Trial Comparing the C-MAC D-Blade Versus the GlideScope in a Mixed Provider and Diverse Patient Population. Anesth Analg. 2016 Mar;122(3):740-750. doi: 10.1213/ANE.0000000000001084. PMID 26579847
- [Background] Ruetzler K, Imach S, Weiss M, Haas T, Schmidt AR. [Comparison of five video laryngoscopes and conventional direct laryngoscopy : Investigations on simple and simulated difficult airways on the intubation trainer]. Anaesthesist. 2015 Jul;64(7):513-9. doi: 10.1007/s00101-015-0051-5. Epub 2015 Jul 15. German. PMID 26174747
- [Background] Piepho T, Weinert K, Heid FM, Werner C, Noppens RR. Comparison of the McGrath(R) Series 5 and GlideScope(R) Ranger with the Macintosh laryngoscope by paramedics. Scand J Trauma Resusc Emerg Med. 2011 Jan 17;19(1):4. doi: 10.1186/1757-7241-19-4. PMID 21241469
- [Background] Al-Ghamdi AA, El Tahan MR, Khidr AM. Comparison of the Macintosh, GlideScope(R), Airtraq(R), and King Vision laryngoscopes in routine airway management. Minerva Anestesiol. 2016 Dec;82(12):1278-1287. Epub 2016 Apr 22. PMID 27103030
- [Background] Maharaj CH, McDonnell JG, Harte BH, Laffey JG. A comparison of direct and indirect laryngoscopes and the ILMA in novice users: a manikin study. Anaesthesia. 2007 Nov;62(11):1161-6. doi: 10.1111/j.1365-2044.2007.05216.x. PMID 17924898
- [Background] El-Tahan MR, Al'ghamdi AA, Khidr AM, Gaarour IS. Comparison of three videolaryngoscopes for double-lumen tubes intubation in simulated easy and difficult airways: a randomized trial. Minerva Anestesiol. 2016 Oct;82(10):1050-1058. Epub 2016 May 12. PMID 27171733